CLINICAL TRIAL: NCT07087574
Title: 3D Printers for Autonomy in the Care of Inpatients in Continuing and Rehabilitation Care
Acronym: AUTARI-3D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-CHITS-011; 2023-A02040-45 (Other: IdRCB)
Record Dates: First submitted 2025-07-09; First posted 2025-07-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Neuro-Degenerative Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient hospitalized in Continuing Care and Rehabilitation Unit (Experimental): Patient suffering from a neurodegenerative disease. Mini Mental Test > 15 and "Eating" criterion of the Katz scale score ≥ 3
  Interventions: Device: adapted cutlery handle printed with 3D printer

INTERVENTIONS:
Device: adapted cutlery handle printed with 3D printer — The patient's autonomy will be assessed by the same ergotherapist, and the quantity of food ingested will be measured by a dietician at 3 similar lunch times:
  * before using the adapted cutlery handles (Day0);
  * when the adapted cutlery handles are used for the first time (Day1);
  * after 3 days' use of the adapted cutlery handles (Day3) On Day0 and Day3, the ergotherapist will carry out an ecological assessment of the meals. Ecological assessment is used in occupational therapy to observe and analyze the patient's interactions with his environment and their repercussions on his ability to perform a task. The aim here is to assess whether the patient exhibits compensation of the upper limb (such as shoulder elevation or trunk inclination) during the meal performed without technical aids (Day0) and that performed after the learning phase of using the adapted handle (Day3).
  The patient's participation will end at the end of the Day3 assessments.

SUMMARY:
Patients hospitalized in Continuing and Rehabilitation Care Units (CRCU) are for the most part elderly people suffering from neurodegenerative diseases, requiring individual, personalized rehabilitation care.

Some of these patients require ergotherapy to help them regain functional ability in everyday activities. The ergotherapist organizes therapeutic activities tailored to patients' needs, with a view to optimizing their level of autonomy.

Loss of autonomy is closely linked to nutritional status, which often tends towards malnutrition in patients admitted to CRCU, with deleterious consequences for the elderly. The use of technical aids to facilitate meal-taking could be a way of alleviating undernutrition. A technical aid is defined as a material aid that enables elderly or disabled people to compensate for a limitation in activity.

The investigators are interested in the use of adapted cutlery, as patients often find it difficult to eat on their own, being unable to grip their cutlery correctly. Commercially adapted cutlery exists, but it is expensive and difficult to use because it is not adapted to each patient (standard size) and is too heavy. What's more, the investigators observe that their use does not necessarily improve the patient's degree of dependence, generally measured by the Katz scale.

The idea of the team of ergotherapist is to offer ergonomic cutlery handles with diameters adapted to patients' degree of prehension. They offer handles with diameters of 25 mm, 30 mm, 35 mm and 40 mm. The diameter is customized according to the hand's flexion capacity, as assessed by a joint and functional assessment. What's original about these technical aids is that they are designed from thermoformable materials with the help of a 3 Dimension printer and Computer-Aided Design and Manufacturing software, in partnership with the Fablab (Fabrication laboratory) in Toulon and the Hyères media library. They have the added advantage of being lightweight and inexpensive.

DETAILED DESCRIPTION:
Patients hospitalized in CRCU will be informed of the research. Those who do not object to participating in the research and who meet the eligibility criteria will be included.

Their participation will begin with an initial functional and joint assessment of the patient's hand by an occupational therapist to determine the diameter of cutlery handles best suited to the patient's grip (25, 30, 35 or 40 mm).

The patient's autonomy ("Eating" criterion on the Katz scale) will be assessed by the same ergotherapist, and the quantity of food ingested will be measured by a dietician at 3 points:

* During a lunch before using the adapted cutlery handles (Day0);
* At lunch when the adapted cutlery handles are used for the first time (Day1);
* At lunch after 3 days' use of the adapted cutlery handles (Day3), corresponding to the learning phase in the use of the technical aid.

Lunches will be similar over the 3 days. These are standard lunches predefined by the unit's dietician.

On Day0 and Day3, the ergotherapist will carry out an ecological assessment of meals. Ecological assessment is used in ergotherapy to observe and analyze the patient's interactions with his environment and their repercussions on his ability to perform a task. The aim here is to assess whether the patient exhibits compensation of the upper limb (such as shoulder elevation or trunk inclination) during the meal performed without technical aids (Day0) and that performed after the learning phase of using the adapted handle (Day3).

The patient's participation will end at the end of the Day3 assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Patient hospitalized in a Continuing Care and Rehabilitation department ;
2. Patient suffering from a neurodegenerative disease (Mini Mental Test score > 15);
3. Age ≥ 18 years;
4. Patient with a score ≥ 3 on the "Eating" criterion of the Katz scale (corresponding to the need for at least partial assistance with meals).

Exclusion Criteria:

1. Opposition of the patient or his relatives to participating in the research ;
2. Patient unable to use hands to eat (amputation, paralysis, etc.);
3. Patient under court protection;
4. Pregnant, parturient or breast-feeding woman;
5. Any other reason which, in the opinion of the investigator, could interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Patients' food autonomy | Day 1
  Eating autonomy is defined by a composite criterion that simultaneously takes into account the following 2 criteria: improvement in the Eating criterion of the Katz scale and the variation in the rate of ingesta with conventional cutlery at Day 0, then on first use of adapted ergonomic cutlery at Day 1. The Eating criterion of the Katz scale comprises four levels, scored from 1 to 4. The higher the score, the greater the need for assistance. Only patients with a score greater than or equal to 3 will be included in this research. The use of ergonomic cutlery handles customized and individualized for food autonomy, will be defined as A SUCCESS, if the patient presents an improvement in the Eating criterion of the Katz scale; accompanied by a rate of ingesta at Day 1 not significantly lower than at Day 0 or a stabilization of the Eating criterion of the Katz scale; accompanied by a rate of ingesta at D1 significantly higher than at D0. A FAILURE, if the patient is in any other situation.

SECONDARY OUTCOMES:
Patients' food autonomy | Day 3
  Patients' food autonomy will be assessed by the same composite criterion defined for the main objective (SUCCES/ECHEC) during a typical lunch, before using the ergonomic cutlery handles (Day 0) and after three days of use (Day 3)
Amount of food ingested | Day 3
  The rate of ingesta over a typical lunch will be quantified by weighing each patient's food before and after meals on Day 0, Day 1 and Day 3. These weighings will be used to calculate the percentage of food ingested during the meal.
Autonomy in food intake ("Eating" criterion) | Day 3
  Patients' autonomy in food intake will be assessed by the "Eating" criterion of the Katz scale during a typical lunch at Day 0, Day 1 and Day 3.The Eating criterion of the Katz scale comprises four levels, scored from 1 to 4. The higher the score, the greater the need for assistance.
Compensations with the upper limb | Day 3
  The presence or absence of compensation with the upper limb at mealtimes will be assessed by an occupational therapist (ecological assessment) with conventional cutlery at Day 0, and after three days' use of ergonomic cutlery handles at Day 3.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Brocandel, Study Director — Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer
Locations (2):
- France (2):
  - SSR Pierre Chevalier, Hyères, Var
  - Hôpital Georges Clemenceau, La Garde, Var

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee KH, Kim DK, Cha YH, Kwon JY, Kim DH, Kim SJ. Personalized assistive device manufactured by 3D modelling and printing techniques. Disabil Rehabil Assist Technol. 2019 Jul;14(5):526-531. doi: 10.1080/17483107.2018.1494217. Epub 2018 Oct 14. PMID 30318956
- [Background] Thorsen R, Cugnod D, Ramella M, Converti R, Ferrarin M. A parametric 3D printed assistive device for people with cerebral palsy - assessment of outcomes and comparison with a commercial counterpart. Assist Technol. 2024 Jan 2;36(1):16-21. doi: 10.1080/10400435.2023.2202696. Epub 2023 May 22. PMID 37083458
- [Background] Katz S, Downs TD, Cash HR, Grotz RC. Progress in development of the index of ADL. Gerontologist. 1970 Spring;10(1):20-30. doi: 10.1093/geront/10.1_part_1.20. No abstract available. PMID 5420677
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- See also: Related Info — https://sante.gouv.fr/soins-et-maladies/prises-en-charge-specialisees/ssr/article/tout-savoir-sur-les-soins-de-suite-et-de-readaptation-ssr
- See also: Related Info — https://www.tutelaire.fr/conseils-et-prevention/tout-savoir-sur-les-ssr-soins-de-suite-et-de-readaptation
- See also: Related Info — https://anfe.fr/qu_est_ce_que_l_ergotherapie/
- See also: Related Info — https://www.ch4v.fr/convalescence-et-readaptation/lactivite-de-reeducation-dans-le-service-de-ssr/
- See also: Related Info — https://www.cairn.info/revue-gerontologie-et-societe1-2010-3-page-157.htm
- See also: Related Info — https://abonnes.hospimedia.fr/articles/20210216-equipement-le-25e-rehab-lab-de-france-ouvre?utm_source=https://www.hospimedia.fr/actualite/articles/20210216-equipement-le-25e-rehab-lab-de-france-ouvre&utm_medium=publicsite&utm_campaign=redirection&utm_term=logged
- See also: Related Info — https://www.otdude.com/ot-practice/3d-printing-applications-for-occupational-therapy-practice/
- See also: Related Info — https://anfe.fr/wp-content/uploads/2022/10/MEMOIRE-IFET-2022-BUROCHAIN-IMPRESSION-3D-IDENTITE-PROFESSIONNELLE-RESILIENCE-f8792a8a.pdf
- See also: Related Info — https://dumas.ccsd.cnrs.fr/dumas-01650672
- See also: Related Info — https://www.estrepublicain.fr/sante/2021/02/10/une-imprimante-3d-au-service-de-la-reeducation-au-centre-bretegnier